CLINICAL TRIAL: NCT04646070
Title: Superomedial Pedicle Versus Inferior Pedicle Techniques in Wise Pattern Reduction Mammaplasty :A Comparison Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Rami Ali Abdelkareem Eleiba, Resident of plastic surgery, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Reduction mammaplasty
Record Dates: First submitted 2020-11-21; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: To Compare Complications of Both Techniques in Wise Pattern Reduction Mammaplasty and to Correlate Between Complications and Patient Mediated Factors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wise pattern reduction mammaplasty using Inferior pedicle (Active Comparator): Wise pattern reduction mammaplasty using Inferior pedicle
  Interventions: Procedure: Reduction mammaplasty
- Wise pattern reduction mammaplasty using superomedial pedicle (Active Comparator)
  Interventions: Procedure: Reduction mammaplasty

INTERVENTIONS:
Procedure: Reduction mammaplasty — Breast reduction surgery
  Other Names: Superomedial pedicle versus Inferior pedicle techniques in wise pattern reduction mammaplasty

SUMMARY:
A comparison study between superomedial and Inferior pedicle techniques in wise pattern reduction mammaplasty

DETAILED DESCRIPTION:
To compare complications of both techniques in wise pattern reduction mammaplasty and to correlate between complications and patient mediated factors

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* previous extensive breast surgery Breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Healthy female patients with macromastia
Enrollment: 30 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-01-20 (Estimated); Study Completion 2021-01-20 (Estimated)

PRIMARY OUTCOMES:
To compare complications of both techniques including nipple areola complex necrosis | 30 days postoperative
  Complications include NAC necrosis and other minor complications including wound dehiscence and seroma or hematoma

SECONDARY OUTCOMES:
To correlate between complications and patient mediated factors | 30 days postoperative
  Patient mediated factors including age, BMI, preoperative hb, suprasternal notch to nipple distance

CONTACTS AND LOCATIONS:
Overall Officials: Safwat Adel hegazy, MD, Study Director — Kafr Elsheikh University
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP